CLINICAL TRIAL: NCT00115193
Title: A Multicenter, Double-Blind, Randomized Study of Pegfilgrastim Administered on the Same Day or the Next Day of R-Chop Chemotherapy in Subjects With Non-Hodgkin's Lymphoma
Brief Title: Pegfilgrastim Administered on the Same Day as Chemotherapy in Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20020134; NCT00066833 (obsolete NCT alias)
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Oncology; NHL; Mantle cell; Diffuse large B-cell; Chemotherapy; RCHOP; Neulasta®; Neutropenia; Pegfilgrastim; Amgen
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neoplasms; Neutropenia | interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Pegfilgrastim
  Interventions: Drug: pegfilgrastim
- Arm B (Active Comparator): Pegfilgrastim
  Interventions: Drug: pegfilgrastim

INTERVENTIONS:
Drug: pegfilgrastim — pegfilgrastim 6 mg on day 1 of each cycle (within 4 hours of chemotherapy completion)
  Arms: Arm A
Drug: pegfilgrastim — pegfilgrastim 6 mg on day 2 of each cycle (at least 24 hours after chemotherapy completion)
  Arms: Arm B

SUMMARY:
The purpose of this study is to provide data on the safety and efficacy of pegfilgrastim when administered on the same day versus the next day of chemotherapy, as measured by the duration of grade 4 neutropenia.

DETAILED DESCRIPTION:
This was a multicenter, double-blind, randomized, phase 2 study of pegfilgrastim given either the same day as or the day after a chemotherapy regimen consisting of cyclophosphamide, doxorubicin, vincristine, prednisone, and rituximab (R-CHOP).

Chemotherapy was administered every 21 days for up to 6 cycles in subjects with aggressive non-Hodgkin's lymphoma (NHL; mantle cell or diffuse large B-cell lymphoma). Subjects were administered R-CHOP on day 1 of each cycle. All subjects were randomized to 1 of 2 treatment arms: arm A subjects were administered pegfilgrastim 6 mg on day 1 of each cycle (within 4 hours of chemotherapy completion); arm B subjects were administered pegfilgrastim 6 mg on day 2 of each cycle (at least 24 hours after chemotherapy completion). All subjects were administered placebo on the day they did not receive pegfilgrastim. A total of 77 subjects were enrolled at 24 centers across the US. Protocol treatment duration for subjects was up to 18 weeks (6 three-week cycles).

ELIGIBILITY:
Inclusion Criteria: - Histologically proven mantle cell lymphoma or histologically proven diffuse large B-cell non-Hodgkin's lymphoma (NHL) according to the REAL classification - Measurable and/or evaluable disease - Previously untreated patients Exclusion Criteria: - Burkitt's or B-lymphoblastic lymphoma - Central nervous system (CNS) involvement - Active infection requiring treatment with systemic anti-infectives within 72 hours of chemotherapy - Prior malignancy within the last 5 years - T-cell lymphoma or history of indolent lymphoma - Prior bone marrow or stem cell transplantation - Known sensitivity to E. coli derived drug products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2003-02; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Reduce the duration of neutropenia and incidence of febrile neutropenia. | The primary outcome will be evaluated at the end of the study.

SECONDARY OUTCOMES:
On the same day as chemotherapy as measured by the incidence of hematologic and non-hematologic toxicities, the number of subjects who received planned doses of chemotherapy on time and response rates. | The secondary outcome will be evaluated at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_11_GCSFSD01_20020134.pdf
- See also: FDA-approved Drug Labeling — http://www.neulasta.com/